CLINICAL TRIAL: NCT02566694
Title: Analysis of Specimens From Patients With Orthopaedic Implants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal National Orthopaedic Hospital NHS Trust (Other)
Collaborators: Massachusetts General Hospital (Other); Coxa, Hospital for Joint Replacement (Other)
Responsible Party: Principal Investigator, Professor Alister Hart, Professor of Orthopaedics, Royal National Orthopaedic Hospital NHS Trust
Other Study IDs: RNOH LIRC
Record Dates: First submitted 2015-09-30; First posted 2015-10-02 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Implants
MeSH Terms: interventions — Drug Implants

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Periprosthetic tissue samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Failed implants: All patients undergoing revision of an orthopaedic implant (previously this was limited to metal hips but this has now expanded to other orthopaedic implants)
  Interventions: Procedure: Implant
- Controls with different failure modes: We will compare findings with different types of orthopaedic implants and categories of failure mode.
  Interventions: Procedure: Implant

INTERVENTIONS:
Procedure: Implant — orthopaedic implant

SUMMARY:
The investigators aim to determine the cause of failure of orthopaedic implants using multi-disciplinary analysis of data from patients who have undergone revision.

DETAILED DESCRIPTION:
The following tests will then be arranged:

* Tribological assessment. The investigators will measure the wear of the explants using: 1) 'out of roundness'; and 2) Coordinate measuring. Semi-quantitative assessment of damage to the explants will also be conducted
* Histological assessment. Tissue sent in formalin may determine the biomarker of diagnosis of metal ion synovitis where applicable
* Metal ion measurement in body fluids where applicable (in patients with metal implants)
* Diamond Light Source (this was approved in the 1st amendment). The tests will involve subjecting formalin fixed tissue to the high energy electron beam of the Diamond Light Source
* Destructive testing of the implant is allowed by the patient (after all non-destructive tests have been performed)
* Protein analysis of fluid and tissue if provided
* Titanium levels from blood samples if provided
* Gene expression testing to assess and understand mechanism of inflammation where applicable

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing revision of an orthopaedic implant (previously this was limited to metal hips but this has now expanded to other orthopaedic implants)

Exclusion Criteria:

* Patients not consenting to the study

Ages: 11 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be both male and female, aged between 11-70 years.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Cause of failure | At time of failure which is likely to be an average of 5 years post operative

CONTACTS AND LOCATIONS:
Overall Officials: Alister Hart, FRCSG(Orth), Principal Investigator — RNOH
Locations (1):
- Royal National Orthopaedic Hospital, Stanmore, London, United Kingdom